CLINICAL TRIAL: NCT00295828
Title: A Pilot Study for the Treatment of Iris Neovascularization With Macugen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hermann Eye Center (Other)
Collaborators: Eyetech Pharmaceuticals (Industry)
Responsible Party: Robert M. Feldman, MD, Hermann Eye Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEF-0510
Record Dates: First submitted 2006-02-22; First posted 2006-02-24 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Iris Neovascularization; Diabetic Retinopathy
Keywords: VEGF; iris neovascularization; diabetic retinopathy; Macugen
MeSH Terms: conditions — Diabetic Retinopathy | interventions — pegaptanib

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Panretinal Photocoagulation (PRP)
  Interventions: Procedure: Panretinal Photocoagulation (PRP)
- 2 (Active Comparator): Panretinal Photocoagulation and Macugen Intravitreal Injection
  Interventions: Other: Pegaptanib Sodium Injection/Panretinal Photocoagulation

INTERVENTIONS:
Other: Pegaptanib Sodium Injection/Panretinal Photocoagulation — Pegaptanib Sodium Injection is a single dose prefilled syringe and is formulated as a 3.47 mg/mL solution. Combined with an ocular laser procedure.
  Other Names: Macugen
  Arms: 2
Procedure: Panretinal Photocoagulation (PRP) — Ocular Laser Procedure
  Other Names: PRP
  Arms: 1

SUMMARY:
The purpose of this study is to determine if a drug called Macugen may help to stop the growth of abnormal blood vessels on the iris that has occurred in the eye(s) as part of diabetic retinopathy.

DETAILED DESCRIPTION:
Diabetic retinopathy is an eye condition caused by diabetes in which new blood vessels grow on the retina (the back, inside part of the eye) and the iris. These vessels are not normal and may leak or break, causing bleeding in the eye. This process can lead to vision loss or blindness, glaucoma (disease of the eye where eye pressures are usually too high resulting in damage to the optic nerve), or other eye problems. This study is to determine if a drug called Macugen may help to stop the growth of these abnormal blood vessels on the iris.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, at least 18 years of age
2. Diabetic retinopathy with iris neovascularization
3. Visual acuity must be light perception or better in the study eye
4. Female patients of childbearing potential must have a negative urine pregnancy test at the screening visit.
5. Written informed consent has been obtained
6. Written authorization for use and release of health and research study information has been obtained

Exclusion criteria:

1. Neovascular glaucoma ( a difficult form of glaucoma to control that leads to a painful eye with high intraocular pressure, corneal swelling, and "cell and flare" in the anterior chamber. Caused by abnormal new blood vessel formation (neovascularization) on the iris, that extends over trabecular meshwork causing closure of angle drainage structures).
2. No light perception in the study eye.
3. Inadequate view of retina for PRP/angiography
4. Anterior chamber intraocular lens implant
5. PRP treatment in the past 60 days. Patients may participate if the PRP treatment is beyond 60 days and has newly diagnosed NVI or has nonregression of previously diagnosed NVI.
6. Previous or current Macugen use
7. Any active ocular infection
8. Any conditions which precludes patients ability to comply with study requirements including completion of the study
9. Female patients who are pregnant, nursing, or planning pregnancy, or who are of childbearing potential and not using a reliable means of contraception
10. Current enrollment in an investigational drug or device study or participation in such a study within 30 days prior to screening
11. Patient has a condition or is in a situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results or may interfere significantly with the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Regression of iris neovascularization and prevention of development of neovascular glaucoma | prospective

SECONDARY OUTCOMES:
Iris angiogram - conducted at screening/treatment visit,week 1, week 3, week 6, week 9, week 12, week 15, week 18, and week 52. | prospective
Regression will be determined by lack of leakage and/or lack of flow through the abnormal vessels. | prospective
Assessment of retina with dilated fundus examination for signs of neovascularization in posterior segment at each follow-up visit | prospective
The complete resolution of iris neovascularization, or regression to less than 2 clock hours of iris neovascularization. | prospective
A clinically significant reduction in the clock hours of angle neovascularization. | prospective
Development of neovascular glaucoma. | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Feldman, MD, Principal Investigator — Hermann Eye Fund & University of Texas -- Houston
Locations (1):
- Robert Cizik Eye Clinic, Houston, Texas, United States